CLINICAL TRIAL: NCT06776133
Title: Evaluation of the Correlation Between Vein Size Inferior Cava and Right Atrial Pressure in Pediatric Age and Creation of a Possible Predictive Model
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PED-RAP-IVC
Record Dates: First submitted 2024-12-03; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-11

CONDITIONS: Congenital Heart Disease; Acquired Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to demonstrate the presence of a correlation between echographic measurements of the inferior vena cava (IVC) normalized for the pediatric population and right atrial pressures (RAP) measured by central venous catheter (CVC) so as to create a predictive model of the value of right atrial pressures using echocardiographic parameters in the pediatric population. This study is single-center longitudinal and involves retrospective and prospective data collection.

DETAILED DESCRIPTION:
Primary objective:

- To build a mathematical predictive model of RAP specifically for paediatric patients from echocardiographic parameters analysed on a retrospective cohort.

Secondary objectives:

* To evaluate the accuracy on the paediatric patient of the mathematical model in use for the estimation of RAP in adult patients in a prospective cohort.
* To test the mathematical model built in this study in a prospective cohort of patients OUTCOME With regard to the primary objective, a new patient-specific model will be built paediatric patient from different methods of ultrasound measurement of the IVC (maximum and minimum diameter expressed as z-score, ratio between the two diameters, ratio between maximum diameter and systolic diameter of the aorta).

systolic diameter of the aorta), as well as the patient's auxo-anthropometric values collected by means of the retrospective data.

With regard to secondary objectives, the mathematical model in use for the patient will be applied adult patient to estimate the RAP in our patients and the value obtained will be compared with the value measured.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 0-18 years undergoing central venous catheter (CVC) placement in the course of the diagnosis performed at our center
* Obtaining informed consent from parent/guardian in case of minors

Exclusion Criteria:

- Patients with univentricular cardiac physiology, nonsinus heart rhythm, mechanical ventilation, Inferior vena cava thrombosis and patients with isomerism

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The retrospective population consists of all patients admitted at the Pediatric Cardiology Unit of IRCCS AOU of Bologna and underwent central venous catheter placement (CVC) during the normal diagnostic-therapeutic course from 1st January of 2012 for which a complete echocardiography was performed within 1 hour of RAP (right atrial pressure) measurement. The prospective population consists of all patients admitted at the Pediatric Cardiology Unit of the IRCCS AOU of Bologna from the time of approval by the ethics committee and undergoing central venous catheter placement for 12 months after the start of this study.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Construction of a mathematical predictive model of RAP specifically for pediatric patients | Once
  The following echocardiographic parameters related to inferior vena cava (IVC) measurements will be analyzed: maximum and minimum expressed as z-score, ratio of the two diameters, ratio of maximum diameter to the systolic systolic aorta. The patient's auxo-anthropometric values collected through the data will also be considered retrospective.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Bonetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy